CLINICAL TRIAL: NCT05268003
Title: A Phase II Study of the Combination of Ponatinib With Mini-hyper CVD Chemotherapy and Venetoclax in Patients With Relapsed or Refractory T-cell Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0802; NCI-2022-01686 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-02-17; First posted 2022-03-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia; Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — ponatinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ponatinib (Experimental): Participants will receive ponatinib (45mg daily) as a single agent for 3 days. These will be called Days -3, -2 and -1
  Interventions: Drug: Ponatinib
- Venetoclax (Experimental): Patients will continue venetoclax 400mg daily on days 1-14 of each 28-day cycle.
  Interventions: Drug: Venetoclax
- Mini-hyper-CVD (Experimental): Chemotherapy will be administered in the inpatient setting, starting on day 1 of each of the cycles 2-8.
  Interventions: Drug: Mini-hyper CVD

INTERVENTIONS:
Drug: Ponatinib — Given by PO
  Arms: Ponatinib
Drug: Venetoclax — Given by PO
  Arms: Venetoclax
Drug: Mini-hyper CVD — Given by IV (vein)
  Arms: Mini-hyper-CVD

SUMMARY:
The addition of ponatinib to mini-hyper-CVD chemotherapy and venetoclax will improve the complete remission rate in patients with relapsed or refractory T-cell acute lymphoblastic leukemia

DETAILED DESCRIPTION:
OBJECTIVES

The addition of ponatinib to mini-hyper-CVD chemotherapy and venetoclax will improve the complete remission rate in patients with relapsed or refractory T-cell acute lymphoblastic leukemia.

Primary Objective:

To assess complete remission (CR) / CR with incomplete count recovery (CRi) rate with the combination of Ponatinib and mini-hyper-CVD chemotherapy and venetoclax.

Secondary Objectives:

To assess the safety of the regimen To assess rate of measurable residual disease (MRD) negative remission To assess duration of response (DOR), progression-free survival (PFS) and overall survival (OS)

Exploratory Objectives:

To assess the level of phospho-LCK in pretreatment samples and correlation with the To assess expression of BCL-2 family proteins

ELIGIBILITY:
Inclusion Criteria:

1. Participants with relapsed or refractory T-cell acute lymphoblastic leukemia defined as receiving one or more cytotoxic containing regimens and A. Bone marrow involvement with ≥ 5% lymphoblasts B. Age ≥ 12 Years and greater than 40kg
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
3. Adequate organ function

   * Serum total bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN for participants with Gilbert's disease
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x ULN, unless clearly due to disease involvement
   * Creatinine clearance ≥50 mL/min (calculated according to institutional standards or using Cockcroft-Gault or Modification of Diet in Renal Disease (MDRD) formula)
4. Women of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use an effective contraception method during the study and for 30 days following the last dose of study drug. Women of non- childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Men who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
5. Participants must provide written informed consent

Exclusion Criteria:

1. Participant is pregnant or breastfeeding
2. Participants under 40kg
3. Participants with uncontrolled active infection
4. Hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
5. Major surgery or radiation therapy within 4 weeks prior to the first study dose
6. Systemic chemotherapy/radiotherapy/investigational therapy within 14 days (with the exception of hydroxyurea, dexamethasone, or one dose of cytarabine) prior to starting therapy
7. No clinical, radiological or laboratory evidence of pancreatitis, including:

   1. Serum lipase must be <2 times the ULN, and
   2. Serum amylase must be <2 times the ULN
8. Symptomatic or untreated leptomeningeal disease or spinal cord compression. Participants with prior h/o CNS disease are eligible as long as no active CNS disease as documented by recent CSF analysis and/or imaging studies.
9. Participants with active heart disease [New York Heart Association (NYHA) class 3-4 as assessed by history and physical examination, unstable angina/stroke/myocardial infarction within the last 6 months]
10. Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

    * Myocardial infarction (MI), stroke, revascularization, unstable angina or transient ischemic attack within 6 months
    * Left ventricular ejection fraction (LVEF) less than 50%
    * Diagnosed or suspected congenital long QT syndrome
    * Clinically significant atrial or ventricular arrhythmias (such as uncontrolled, clinically significant atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) as determined by the treating physician
    * Prolonged QTc interval on pre-entry electrocardiogram (> 480 msec) unless corrected after electrolyte replacement or Currently taking drugs that are known to have a risk of causing prolonged QTc or torsades de pointes (TdP) (unless these can be changed to acceptable alternatives or discontinued)
    * History of venous thromboembolism including deep venous thrombosis or pulmonary embolism within the past 3 months, excluding line-associated DVT of the upper extremity
    * Uncontrolled hypertension (diastolic blood pressure >100mmHg; systolic >150mmHg).

10. Uncontrolled hypertriglyceridemia (triglycerides > 450mg/dL) 11. History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years. Participants with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses) 12. Taking any medications or herbal supplements that are known to be strong inhibitors (such as fluconazole, ketoconazole, voriconazole, and clarithromycin) or inducers (such as rifampin, rifabutin, phenytoin, carbamazepine, and St. John's Wort) of cytochrome P450 (CYP)3A4 within at least 7 days before the first dose of ponatinib or within 3 days of starting venetoclax.

13. Consumed grapefruit, grapefruit products, Seville oranges, or star fruit within 3 days prior to starting venetoclax 14. Malabsorption syndrome or other conditions that preclude enteral route of administration 15. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the participants inappropriate for enrollment into this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
To determine the complete remission (CR) / CR with incomplete count recovery (CRi) rate with the combination of Ponatinib and mini-hyper-CVD chemotherapy and venetoclax. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jain Nitin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05268003/ICF_000.pdf